CLINICAL TRIAL: NCT02134808
Title: Placebo-Controlled Trial of Creatine Augmentation for Adolescent Females With Treatment-Resistant Major Depressive Disorder: a Magnetic Resonance Spectroscopy Study
Brief Title: Creatine Augmentation for Adolescent Females With Treatment-Resistant Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Perry Renshaw (Other)
Responsible Party: Sponsor-Investigator, Perry Renshaw, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00073442
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Creatine; Brain Chemistry; Magnetic Resonance Spectroscopy; Treatment Resistance; Selective Serotonin Reuptake Inhibitor (SSRI) Resistance
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Creatine (Active Comparator): Subjects randomized to this study arm will receive 10 grams of creatine daily for 8 weeks.
  Interventions: Drug: Creatine
- Placebo (Placebo Comparator): Subjects randomized to this study arm will receive 10 grams of placebo daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Creatine — Creatine is a nutritional supplement.
  Other Names: Creatine Monohydrate
  Arms: Creatine
Drug: Placebo — The placebo is an inactive ingredient similar in appearance, weight and density to the active treatment.
  Other Names: Placebo Control
  Arms: Placebo

SUMMARY:
The primary hypothesis is that compared to placebo, 10g of daily creatine monohydrate for eight weeks will be associated with significant increases in frontal lobe phosphocreatine and beta-nucleoside triphosphate (β-NTP) concentrations. A secondary hypothesis is that decreased depressive symptoms measured with the Children's Depression Rating Scale-Revised (CDRS-R) and Montgomery-Asberg Depression Rating Scale (MADRS) will be reciprocally correlated with increased β-NTP concentrations.

DETAILED DESCRIPTION:
The current protocol seeks to expand upon the investigators previous work by opening recruitment on a pilot study of creatine 10g daily vs. placebo as a treatment for female adolescents with SSRI-resistant MDD. The purpose of the pilot study is twofold: A) to evaluate several aspects of the feasibility of creatine supplementation as a treatment for this population; and B) to estimate the effect size of adjunctive creatine, to inform the design and implementation of a potential future efficacy trial.

ELIGIBILITY:
MAJOR DEPRESSIVE DISORDER SUBJECTS

Inclusion Criteria:

1. Participants must be female.
2. Participants must be able to grant informed consent (age >18), or parent/guardian permission plus participant assent (age <18).
3. Participants must meet DSM criteria for Major Depressive Disorder (MDD), with current mood state depressed for > 2 weeks.
4. Participants must be between the ages of 12 and 21.
5. Current CDRS-R raw score of > 40 or MADRS score > 25; and CGI-S score > 3.
6. Participants may be enrolled in individual and/or group psychotherapy, if it has been ongoing for at least 8 weeks.
7. Participants must have been in treatment with an SSRI for at least 8 weeks, the last 4 of which were at a dosage of > 20 mg per day of fluoxetine or its equivalent, e.g. 20 mg per day of paroxetine, 20 mg citalopram, 10 mg escitalopram, or 100 mg sertraline. If the participant attempted, but could not tolerate, a dose comparable to 20 mg fluoxetine, they will be considered eligible. (This definition of "Adolescent SSRI Resistant Depression" is modified from the NIH-sponsored, $17 million TORDIA Randomized Controlled Trial [http://clinicaltrials.gov/ct2/show/NCT00018902].

Exclusion Criteria:

1. Unstable co-morbid medical, neurological, or psychiatric disorder.
2. Current DSM criteria for substance abuse or dependence (excepting nicotine/cigarettes).
3. Clinically significant suicidal or homicidal risk.
4. Pre-existing renal disease.
5. Proteinuria on baseline urinalysis testing.
6. Pregnancy or breastfeeding.
7. Sexually active and unwilling to practice contraception during the study.
8. Contraindication to magnetic resonance imaging (e.g. ferromagnetic implant or claustrophobic anxiety).
9. History of hypersensitivity to creatine.
10. History of a previous failed therapeutic trial of creatine.
11. Participants may be outpatients or inpatients, but incarcerated persons will be excluded because this study is not approved for "Research Involving Prisoners."

Study Withdrawal Criteria:

1. Withdrawal of parental permission, participant informed consent or participant assent.
2. Onset of a psychotic disorder or bipolar disorder.
3. Intolerable, or clinically-significant side effects to creatine.
4. Worsening depression, as demonstrated by an increase in CDRS-R or MADRS score > 25% from baseline.
5. Positive pregnancy test.
6. A significant change to the participant's medication or psychotherapy treatment from the regimen reported at their baseline/screening visit (e.g. if the SSRI is discontinued).
7. Incarceration, as the study is not approved to conduct "Research Involving Prisoners."
8. If a clinically-significant intracranial lesion is found by the Radiologist on a participant's baseline brain scan, they will be withdrawn from the study and referred for appropriate medical care.
9. The principal investigator retains the right to withdraw participants from the study without their permission, in the event they are unwilling or unable to maintain adherence with the research protocol.

HEALTHY COMPARISON SUBJECTS

Inclusion Criteria:

1. Participants must be able to grant informed consent (age > 18), or parent/guardian permission plus participant assent (age < 18).
2. Participants must be female.
3. Participants must be between the ages of 12 and 21 years.
4. Participants must not meet DSM criteria for a current psychiatric illness or substance use disorder.
5. Participants must have a CDRS-R score < 30.

Exclusion Criteria:

1. Unstable medical or neurological illness.
2. Clinically-significant psychiatric or substance use disorder.
3. Pregnant subjects, due to the unknown effects of MRI/MRS scans on a fetus. In addition, women of childbearing potential who are unable or unwilling to practice contraception during the study will be excluded. Female participants who are of childbearing potential must have a negative urine pregnancy test before the MRI/MRS scan.
4. Participants with a contraindication to MRI/MRS scanning, such as a metallic implant.

Study Withdrawal Criteria:

1. Withdrawal of parental permission or participant assent.
2. Onset of a psychotic disorder or depression.
3. Positive pregnancy test.
4. A significant change to the participant's medication or psychotherapy treatment from the regimen reported at their baseline/screening visit, unless directed by the principal investigator.

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kondo, MD, Study Director — University of Utah; Perry F Renshaw, MD, PhD, MBA, Principal Investigator — University of Utah
Locations (1):
- University of Utah School of Medicine, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kondo DG, Sung YH, Hellem TL, Fiedler KK, Shi X, Jeong EK, Renshaw PF. Open-label adjunctive creatine for female adolescents with SSRI-resistant major depressive disorder: a 31-phosphorus magnetic resonance spectroscopy study. J Affect Disord. 2011 Dec;135(1-3):354-61. doi: 10.1016/j.jad.2011.07.010. Epub 2011 Aug 9. PMID 21831448

RESULTS

PARTICIPANT FLOW:
Groups:
- Creatine: 28 Subjects randomized to this study arm will receive 10 grams of creatine daily for 8 weeks.
  Creatine: Creatine is a nutritional supplement.
- Placebo: 23 Subjects randomized to this study arm will receive 10 grams of placebo daily for 8 weeks.
  Placebo: The placebo is an inactive ingredient similar in appearance, weight and density to the active treatment.
- Healthy Comparison: 20 Subjects seen for screening and baseline scan. No randomization or treatment intervention for subjects enrolled as a Healthy Comparison.
Period: Overall Study
Arm/Group | Creatine | Placebo | Healthy Comparison
Started | 28 | 23 | 20
Completed | 24 | 19 | 20
Not Completed | 4 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Participants are assessed using Montgomery-Åsberg Depression Rating Scale (MADRS) and Children's Depression Rating Scale-Revised (CDRS-R).
Groups:
- Total: Total of all reporting groups
Arm/Group | Creatine | Placebo | Healthy Comparison | Total
Number analyzed (Participants) | 28 | 23 | 20 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 9 | 7 | 30
  Between 18 and 65 years | 14 | 14 | 13 | 41
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.6 (2.2) | 17.8 (2.0) | 17.4 (3.2) | 17.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 20 | 71
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 27 | 19 | 16 | 62
  Black or African American | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Hispanic or Latino | 1 | 3 | 1 | 5
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Other | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 23 | 20 | 71

OUTCOME MEASURES:

1. Primary Outcome: Brain Phosphocreatine (PCr) Concentrations
Description: PCr will be measured through phosphorus magnetic resonance spectroscopy (31P-MRS). This will be performed in a 3 Tesla magnetic resonance imaging (MRI) scanner.
  Creatine concentration before and after treatment. By convention, 31P MRS data are typically reported as metabolite ratios.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Creatine: 28 Subjects randomized to this study arm will receive 10 grams of creatine daily for 8 weeks.
- Placebo: 23 Subjects randomized to this study arm will receive 10 grams of placebo daily for 8 weeks.
Arm/Group | Creatine | Placebo | Healthy Comparison
Number analyzed (Participants) | 28 | 23 | 20
Ratio
  Baseline | .1812802 (.011512) | .1796093 (.0070168) | .1850427 (.0059435)
  Week 8 | .1876206 (.0121833) | .181464 (.008267) | NA (NA) — Healthy Comparison participants were only scanned at baseline.

2. Secondary Outcome: Children's Depression Rating Scale-Revised (CDRS-R); Montgomery-Asberg Depression Rating Scale (MADRS)
Description: The Children's Depression Rating Scale-Revised (CDRS-R) and Montgomery-Asberg Depression Rating Scale (MADRS) will be administered to understand the severity of depressive symptoms, and how these symptoms change throughout the course of the study. The CDRS-R has a range of minimum score 17 and maximum score 113, with higher scores indicating more severe depression. The MADRS has a range of 0 to 60 with higher scores indicating more severe depressive symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Creatine | Placebo | Healthy Comparison
Number analyzed (Participants) | 28 | 23 | 20
score on a scale
  CDRS-R Baseline | 58.28571 (6.980699) | 60.3913 (6.719978) | 21.9 (2.425739)
  CDRS-R Week 8 | 41.95833 (12.47773) | 44.15789 (10.25921) | NA (NA) — Healthy Comparison participants were only assessed at baseline.
  MADRS Baseline | 28.71428 (5.394491) | 31.47826 (4.832368) | 2.315789 (2.029029)
  MADRS Week 8 | 16.16667 (11.21981) | 18.73684 (11.29819) | NA (NA) — Healthy Comparison participants were only assessed at baseline.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from participants at every visit, starting after the treatment intervention was dispensed at baseline. Adverse events were assessed up to 8 weeks.
Description: Healthy comparison participants were only seen for a baseline scan. Healthy comparison participants were not exposed to any treatment intervention, therefore, adverse events were not collected.
Arm/Group | Creatine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/28 | 0/23
Other Adverse Events (participants affected / at risk) | 18/28 | 15/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creatine (N=28) | Placebo (N=23)
Suicidal Ideation/Behavior (Psychiatric disorders) | 1 (1) | 0 (0) — A 17 year old participant was hospitalized for a suicide attempt that occurred 5 days after randomization. The participant had a history of four previous suicide attempts. Subsequently, the criteria changed to reduce the risks of participation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Creatine (N=28) | Placebo (N=23)
Abdominal cramp, Nausea, Indigestion, Diarrhea (Gastrointestinal disorders) | 15 (35) | 12 (26)
Headache (Nervous system disorders) | 18 (35) | 15 (37)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 14 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT02134808/Prot_SAP_000.pdf